CLINICAL TRIAL: NCT04841122
Title: Improved Patient Safety for Acute Restless Medical Patients With Supplemental Observation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated after 6 months due to recruitment and data collection challenges.
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Mette Geil Kollerup, Principal investigator and postdoc., Aalborg University Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: N-20200079
Record Dates: First submitted 2021-03-25; First posted 2021-04-12 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camera observation (Active Comparator): Camera observation
  Interventions: Device: Camera observation
- No camera observation (No Intervention): No intervention

INTERVENTIONS:
Device: Camera observation — Supplemental camera observation directly linked to the nurse's phone
  Arms: Camera observation

SUMMARY:
The aim of the study is to investigate whether supplemental camera observation directly linked to the nurse's phone will improve patient safety for acute medical care patients', who are restless, confused or in risk of development of acute delirium. The setting is an acute medical care ward.

The expected result is a reduced incidence of patients with delirious condition, patients who fall or unintentionally remove intravenous access or catheters. Thus, higher patient safety and more efficient patient trajectories are expected, as well as a reduced need for treatment, care and rehabilitation after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age with a CAM score of 2 or higher.

Exclusion Criteria:

* paranoia
* severe dementia
* suicidal
* need for permanent guard

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Confusion Assessment Score | First measurement at admission and second measurement within 24 hours.
  Assessed by Confusion Assessment Method (CAM) screening tool. Minimum value is 0, Maximum value is 4. Higher score means higher risk of developing Delirium.

SECONDARY OUTCOMES:
Number of patient falls | The time the patient is assessed during the observation period.
  Incidence of patient falls observed by the nurse during the observation period.
Discontinuation of accesses | The time the patient is assessed during the observation period.
  Number of patient discontinuation of e.g. oxygen mask, peripheral venous catheter, bladder catheters
Number of administrations of sedatives | The time the patient is assessed during the observation period.
  Number of OR administrations and number of IV administrations (specific sedatives e.g. Methylphenidate, Haloperidol, Midazolam).

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg Universityhospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No